CLINICAL TRIAL: NCT07375654
Title: A Comparative Study on the Efficacy of The Combined Use of Cyclosporine and Metformin in the Treatment of Psoriasis vs Cyclosporine Alone
Brief Title: Combined Use of Cyclosporine and Metformin in Treatment of Psoriasis vs Cyclosporine Alone
Acronym: CsA/Met
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Fahim, Assistant Professor of Dermatology,Faculty of Medicine ,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-308-2024
Record Dates: First submitted 2026-01-07; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
Keywords: psoriasis; cyclosporin; metformin
MeSH Terms: conditions — Psoriasis | interventions — Cyclosporine; Metformin

STUDY DESIGN:
Intervention Model Description: * Patients will be divided randomly (by simple randomization) into 2 equal groups: Group A: (16) patients will receive Cyclosporine (dose 3 mg/kg). And group B: (16) patients will receive Cyclosporine and Metformin (500 mg twice daily).
  * The instruction to the both groups will be identical and they will receive the treatment for a total of 3 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporin (CSA) (Active Comparator): Group A: (16) patients will receive Cyclosporine (dose 3 mg/kg),orally twice per day for 3months
  Interventions: Drug: Cyclosporin (CSA)
- Cyclosporin plus Metformin (Active Comparator): Group B: (16) patients will receive Cyclosporine(3mg/kg/day), orally and Metformin (500 mg twice daily) ,orally for 3 months
  Interventions: Drug: Cyclosporin (CSA); Drug: Metformin (500 mg Twice a day)

INTERVENTIONS:
Drug: Cyclosporin (CSA) — Cyclosporine (dose 3 mg/kg),orally twice per day for 3 months
Drug: Metformin (500 mg Twice a day) — Metformin (500 mg twice daily),orally for 3 months
  Arms: Cyclosporin plus Metformin

SUMMARY:
This study is a comparative clinical study evaluating the efficacy of combined therapy using cyclosporine and metformin versus cyclosporine alone in the treatment of psoriasis. Psoriasis is a chronic inflammatory skin disease that often requires systemic therapy in moderate to severe cases. Cyclosporine is an effective immunosuppressive agent; however, its long-term use is limited by potential adverse effects.

Metformin, a commonly used antidiabetic drug, has shown anti-inflammatory and immunomodulatory properties, which may enhance treatment outcomes in psoriasis. This study aims to assess whether adding metformin to cyclosporine improves clinical response compared to cyclosporine monotherapy.

DETAILED DESCRIPTION:
Psoriasis is a chronic, immune-mediated inflammatory skin disease characterized by erythematous, scaly plaques and a relapsing course. It has a significant negative impact on patients' quality of life and is frequently associated with metabolic comorbidities, including insulin resistance and obesity. Management of moderate to severe psoriasis often requires systemic therapy to achieve adequate disease control.

Cyclosporine is a well-established systemic immunosuppressive drug used in the treatment of moderate to severe psoriasis due to its rapid onset of action and effectiveness in reducing disease severity. Its mechanism involves inhibition of T-cell activation and cytokine production. However, long-term use of cyclosporine is limited by potential adverse effects, particularly nephrotoxicity, hypertension, and metabolic disturbances. Therefore, strategies to enhance its efficacy while potentially allowing dose reduction are of clinical importance.

Metformin is an oral hypoglycemic agent widely used in the management of type 2 diabetes mellitus. Beyond its glucose-lowering effect, metformin has demonstrated anti-inflammatory, immunomodulatory, and antiproliferative properties. Recent evidence suggests that metformin may play a beneficial role in inflammatory and immune-mediated diseases, including psoriasis, through modulation of inflammatory cytokines and improvement of insulin resistance, which is commonly observed in psoriatic patients.

This study is designed as a comparative clinical study to evaluate the efficacy of combined therapy using cyclosporine and metformin versus cyclosporine monotherapy in the treatment of psoriasis. The primary objective is to assess whether the addition of metformin enhances the clinical response compared to cyclosporine alone. Treatment efficacy will be evaluated using standardized clinical assessment tools for psoriasis severity, along with monitoring of treatment safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients of both genders
* Patients clinically diagnosed as moderate to severe psoriasis candidate for systemic treatment with Psoriasis Area Severity Index (PASI >10), Body Surface Area (BSA>10), Dermatology Life Quality Index (DLQI>10).(Laura Salgado-Boquete et al., 2021).
* Patients with new active lesions and also patient with chronic lesions (with periods of remission and exacerbation)

Exclusion Criteria:

* Erythrodermic and pustular psoriasis.
* Patients with systemic illness ( renal, hepatic and uncontrolled hypertension ).
* Pregnant and lactating females.
* Patients receiving systemic treatment relevant to psoriasis within 3 months before enrollment into the study or topical treatment relevant to psoriasis within 1 month before.
* Patients with other dermatological conditions.
* Patients with high uric acid level .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure 1 Change in Psoriasis Area and Severity Index (PASI) | Baseline (Pretreatment) ,Post-treatment(At 3 months),At 6 months
  Comparison of PASI scores before and after treatment within each group and between both treatment groups.
  Unit of Measure:
  PASI score
  Scale:
  0-72 (higher scores indicate more severe psoriasis)
Primary Outcome Measure 2 Change in Body Surface Area (BSA) | Baseline (pretreatment), 3 months, and 6 months post-treatment
  Comparison of the percentage of body surface area affected by psoriasis before and after treatment within each group and between both treatment groups.
  Unit of Measure:
  Percentage of body surface area (%)
  Scale:
  0-100% (higher percentages indicate greater skin involvement)
Primary Outcome Measure 3 Change in Dermatology Life Quality Index (DLQI) | Baseline (pretreatment), 3 months, and 6 months post-treatment
  Comparison of DLQI scores before and after treatment within each group and between both treatment groups.
  Unit of Measure:
  DLQI score
  Scale:
  0-30 (higher scores indicate greater impairment of quality of life)

SECONDARY OUTCOMES:
Patient satisfaction . | Post treatment(AT 3 months)
  Patients' Global Satisfaction Scale ranging from -1 to 3. Patient satisfaction is graded as excellent (3), moderately satisfied (2), poorly satisfied (1), not satisfied (0), or condition worsened (-1), with higher scores indicating greater patient satisfaction and better clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Salah El-Mesidy, Assistant Professor, Principal Investigator — Cairo University; Aya Mohamed Fahim, Assistant Professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code